CLINICAL TRIAL: NCT06714396
Title: A Randomized, Placebo-Controlled, Double-Blind, Single-Dose, Phase 1 Study to Explore the PK/PD Relationship of QRL-101 in People Living With ALS
Brief Title: A Study Exploring the PK/PD Relationship of QRL-101 in Adults With ALS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: QurAlis Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: QRL-101-04
Record Dates: First submitted 2024-11-27; First posted 2024-12-03 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- QRL-101 (Experimental): Single doses of QRL-101 will be orally administered. The dose levels may change subject to available nonclinical, clinical, safety, and PK data.
  Interventions: Drug: QRL-101
- Placebo (Experimental): Single doses of comparator placebo will be orally administered. The dose levels may change subject to available nonclinical, clinical, safety, and PK data.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: QRL-101 — Single doses of QRL-101 will be orally administered. The dose levels may change subject to available nonclinical, clinical, safety, and PK data.
  Arms: QRL-101
Other: Placebo — Single doses of compartor placebo will be orally administered. The dose levels may change subject to available nonclinical, clinical, safety, and PK data.
  Arms: Placebo

SUMMARY:
This Phase 1 randomized, placebo-controlled, double-blind study will evaluate the PK/PD relationship of single doses of QRL-101 in 12 ALS participants. The study will also assess safety and tolerability in participants receiving either QRL-101 or placebo.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, single-dose, single-site, Phase 1 study to explore the pharmacokinetics (PK) and pharmacodynamics (PD) of single doses of QRL-101 in participants with ALS. In addition, the safety and tolerability of QRL-101 will be evaluated. Single doses of QRL-101 or placebo will be administered as an oral liquid to approximately 12 participants with ALS. The study will explore the PK, PD, and PK/PD relationship among three dose levels of QRL-101 and placebo. The randomization will be 1:1:1:1 for the four study groups and will be conducted in 3 blocks (cohorts) of 4, where participants will be randomized 3:1 (QRL-101:placebo) for increasing dose levels of QRL-101.

ELIGIBILITY:
INCLUSION CRITERIA

1. Age 18 to 80 years of age inclusive at the time of signing the informed consent.
2. Diagnosis of ALS, by either Gold Coast Criteria or El Escorial Criteria (possible, probable laboratory supported, probable, or definite)
3. Clinical chemistry laboratory values within acceptable range for the population, as per investigator judgment.
4. Body mass index of 18 to 32 kg/m2 (inclusive).
5. Willing and able to practice effective contraception.

EXCLUSION CRITERIA

1. Currently enrolled in any other clinical trial involving a study drug, off-label drug or device use, or any other type of medical research judged not scientifically or medically compatible with this study.
2. History or presence of medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric, or neurological disease, convulsions, or any clinically significant laboratory abnormality that, in the judgment of the investigator, indicate a medical problem that would preclude study participation.
3. Off-label use of drugs or devices that are being used or investigated as disease-modifying therapies in ALS
4. Participated in another clinical study within 30 days, or 5 half-lives of the previous investigational product, whichever is greater, prior to the planned randomization date.
5. Taking any prescription or nonprescription medicines that are cytochrome P450 3A4 inducers, inhibitors, or substrates within 30 days or 5 half-lives, whichever is greater, prior to the planned randomization date

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2025-08-22 (Actual)

PRIMARY OUTCOMES:
QRL-101 plasma concentration | Baseline through Follow up (Day 10)
PK/PD Relationship: Strength-Duration Time Constant (SDTC) | Baseline through Follow up (Day 10)

SECONDARY OUTCOMES:
Safety and Tolerability: Adverse Events (AEs) | Baseline through Follow up (Day 10)
Safety and Tolerability: Serious Adverse Events (SAEs) | Baseline through Follow up (Day 10)
Plasma PK profile: Maximum concentration observed (Cmax) | Baseline through Follow up (Day 10)
Plasma PK profile: Time of maximum drug concentration (Tmax) | Baseline through Follow up (Day 10)
Plasma PK profile: Area under the concentration time curve from time 0 to 24 hours (AUC0-24hr) | Baseline through Follow up (Day 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands, Netherlands